CLINICAL TRIAL: NCT03249402
Title: An Open-label Drug-drug Interaction Study in Healthy Female Adult Subjects to Investigate the Effect of Multiple Oral Doses of JNJ-42847922 on the Steady-state Pharmacokinetics of an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel
Brief Title: A Study to Evaluate the Effect of Multiple Oral Doses of JNJ-42847922 on the Steady-state Pharmacokinetics of an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel in Healthy Female Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108351; 2016-004725-16 (EudraCT Number); 42847922MDD1003 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination; seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Contraceptive Tablet + JNJ-42847922 (Experimental): All participants will receive one oral contraceptive (OC) tablet containing ethinyl estradiol (EE) 0.03 milligram (mg) and levonorgestrel (LN) 0.15 mg once daily on Days 1 to 21 for both cycle 1 and cycle 2. In addition, in cycle 2, participants will receive 40 mg of JNJ-42847922 once daily on Days 14 to 21. Participants will not be given OC tablet on Days 22 to 28 during cycle 1 and cycle 2 (tablet-free period).
  Interventions: Drug: Ethinyl Estradiol + Levonorgestrel; Drug: JNJ-42847922

INTERVENTIONS:
Drug: Ethinyl Estradiol + Levonorgestrel — Participants will receive one OC tablet containing EE 0.03 mg and LN 0.15 mg once daily on Days 1 to 21 in cycles 1 and 2.
  Other Names: Microgynon 30
Drug: JNJ-42847922 — Participants will receive 40 mg of JNJ-42847922 once daily on Days 14 to 21 in cycle 2.

SUMMARY:
The purpose of this study is to evaluate the effect of multiple 40 milligram (mg) doses of JNJ-42847922 on the steady state pharmacokinetics (PK) of multiple doses of a combination oral contraceptive (OC) containing ethinyl estradiol (EE) and levonorgestrel (LN) in healthy female adult partcipants.

ELIGIBILITY:
Inclusion Criteria:

* Be female of childbearing potential (women with tubal ligation are not accepted)
* Have a body weight equal to or over 45 kilogram (kg) and a body mass index (BMI) 23 within the range of 18 to 30 kilogram / square meter (kg/m^2) inclusive
* Have a systolic blood pressure between 90 and 140 millimeter of mercury (mmHg), inclusive, and diastolic blood pressure no higher than 90 mmHg
* Agree not to donate eggs (ova, oocytes) during the study and for at least 90 days after receiving the last dose of study drug
* Have a negative serum pregnancy test at screening and a negative predose urine pregnancy test on Day1 and Day 21 of Cycle 1 and Cycle 2

Exclusion Criteria:

* Participant has a past history of heart arrhythmias (extrasystolic, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participant is currently pregnant or planning to become pregnant or lactating (from screening through at least 8 weeks after receiving the last dose of study drug)
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody positive, or other clinically active liver disease, or tests positive for HBsAg or hepatitis C virus antibody at screening.
* Participant has a history of or present allergy to the oral contraceptive (OC) or JNJ-42847922, or drugs of these classes, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Participant has a history of alcohol/drug abuse or dependence within 12 months of the study: history of regular alcohol consumption averaging greater than (>) 14 drinks/week for women within 6 months of screening

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) in Cycle 1 | Cycle 1: Predose (Day 21), 30 minute (min), 1 hour (h), 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 20h, 24h, 28h, 36h, 48h and 72h Postdose
  The Cmax is the maximum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) in Cycle 2 | Cycle 2: Predose (Day 21), 30 minute (min), 1 hour (h), 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 20h, 24h, 28h, 36h, 48h and 72h Postdose
  The Cmax is the maximum observed plasma concentration.
Trough Plasma Concentration (Ctrough) in Cycle 1 | Cycle1: Predose (Day 21)
  The (Ctrough) is the observed plasma concentration just prior to the beginning of a dosing interval.
Trough Plasma Concentration (Ctrough) in Cycle 2 | Cycle 2: Predose (Day 21)
  The (Ctrough) is the observed plasma concentration just prior to the beginning of a dosing interval.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) at Cycle 1 | Cycle 1: Predose (Day 21), 30 minute (min), 1 hour (h), 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 20h, Day 22: 24h Postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) at Cycle 2 | Cycle 2: Predose (Day 21), 30 minute (min), 1 hour (h), 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 20h, Day 22: 24h Postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 87 Days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- SGS Life Science Services, Antwerp, Belgium